CLINICAL TRIAL: NCT04146701
Title: Metabolomics and Microbiomics in Cardiovascular Diseases
Acronym: MEMORIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Michael Behnes, Attending physician, adjunct professor, Universitätsmedizin Mannheim
Other Study IDs: 2019-1093N-MA
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Acute Heart Failure; NSTEMI - Non-ST Segment Elevation MI; STEMI - ST Elevation Myocardial Infarction; Myocardial Infarction, Acute; Sepsis; Cardiomyopathies; Dilated Cardiomyopathy; Ischemic Cardiomyopathy
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction; Myocardial Infarction; Sepsis; Cardiomyopathies; Cardiomyopathy, Dilated | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Withdrawl of peripheral venous blood (ca. 40ml) in EDTA, and ammonium heparin serum tubes at the time of acute disease status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Acute heart failure: All consecutive patients admitted with acute heart failure to University Medical Center Mannheim. One venous blood withdraw will be performed. Demographic and clinical data will be documented.
  Interventions: Other: Blood draw
- STEMI: All consecutive patients admitted with STEMI to University Medical Center Mannheim. One venous blood withdraw will be performed. Demographic and clinical data will be documented.
  Interventions: Other: Blood draw
- NSTEMI: All consecutive patients admitted with NSTEMI to University Medical Center Mannheim. One venous blood withdraw will be performed. Demographic and clinical data will be documented.
  Interventions: Other: Blood draw
- Ischemic cardiomyopathy: All consecutive patients with an implantable cardioverter defibrillator (ICD) due to ischemic cardiomyopathy and LVEF <35% presenting for ICD check-up to University Medical Center Mannheim. One venous blood withdraw will be performed. Demographic and clinical data will be documented.
  Interventions: Other: Blood draw
- Non-ischemic cardiomyopathy: All consecutive patients with an implantable cardioverter defibrillator (ICD) due to non-ischemic cardiomyopathy and LVEF <35% presenting for ICD check-up to University Medical Center Mannheim. One venous blood withdraw will be performed. Demographic and clinical data will be documented.
  Interventions: Other: Blood draw
- Sepsis: All consecutive patients admitted with sepsis or septic shock to University Medical Center Mannheim. One venous blood withdraw will be performed. Demographic and clinical data will be documented.
  Interventions: Other: Blood draw
- Healthy controls: Clinically inapparent group as controls. One venous blood withdraw will be performed. Demographic and clinical data will be documented.
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — venous blood withdraw (ca. 40ml)

SUMMARY:
"MEtabolomics and MicrObiomics in caRdIovAscular diseases Mannheim (MEMORIAM) " is a single-center, prospective and observational study investigating to identify disease-specific metabolic, respectively microbiomic, patterns of patients with high-risk cardiovascular diseases. High-risk cardiovascular diseases comprise patients suffering from acute heart failure (AHF), ST-segment elevation myocardial infarction (STEMI), non-ST-segment elevation myocardial infarction (NSTEMI), sepsis, septic shock, ischemic and non-ischemic cardiomyopathy.

DETAILED DESCRIPTION:
Scientific evidence about the metabolomic and microbiomic changes in high-risk cardiovascular patients is still lacking.

The acute, critical or progressive disease status predestinies to relevant changes in cardiovascular metobolism. High-risk patients in the present trial comprise those with acute heart failure, myocardial infarction (STEMI and NSTEMI), sepsis, septic shock, ischemic and non-ischemic cardiomyopathy with severely reduced left ventricular ejection fraction (LVEF <35%).

Therfore this study investigates to identify disease-specific patterns of metabolic and microbiomic changes. These patterns may help to understand pathophysiology at the metabolic stages and find out those patients being at highest risk of adverse future outcome.

ELIGIBILITY:
Inclusion Criteria:

* above mentioned diseases, diagnosis according to respective guideline
* written informed consent

Exclusion Criteria:

* under 18 years
* cancer
* rheumatic diseases
* infections (except septic group)
* higher grade heart valve diseases

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suffering from acute cardiovascular diseases such as acute heart failure, STEMI, NSTEMI, ischemic and dilative cardiomyopathies and sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-specific metabolic/microbiomic biomarker patterns. | Within 24h after disease onset
  Expression of disease-specific metabolic/microbiomic biomarker patterns at the time of acute disease presentation

SECONDARY OUTCOMES:
All-cause and cardiovascular mortality. | 12 months after inclusion
  All-cause and cardiovascular mortality, at 6 months and 12 months
Cardiac rehospitalization. | 12 months after inclusion
  Cardiac rehospitalization, at 6 months and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Behnes, PD Dr., Study Director — University Medical Center Mannheim
Locations (1):
- University Medical Center Mannheim, Mannheim, Germany